CLINICAL TRIAL: NCT07269210
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of LY3561774 (Solbinsiran) in Adults With Severe Hypertriglyceridemia
Brief Title: A Study of Solbinsiran (LY3561774) in Participants With Severe Hypertriglyceridemia
Acronym: SOLARIS-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27775; J3F-MC-EZCC (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Severe Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Solbinsiran (Experimental): Participants will receive solbinsiran subcutaneously (SC)
  Interventions: Drug: Solbinsiran
- Placebo (Placebo Comparator): Participants will receive placebo SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solbinsiran — Administered SC
  Other Names: LY3561774
  Arms: Solbinsiran
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of solbinsiran in lowering triglycerides and other lipid measures compared to placebo in participants with severe hypertriglyceridemia. Participants will receive two subcutaneous injections.

ELIGIBILITY:
Inclusion Criteria:

* History of fasting triglyceride levels of ≥500 milligrams per deciliter (mg/dL), based on medical history
* Fasting triglyceride level ≥500 mg/dL at two separate visits during screening (at least 7 days apart)
* Have a body mass index (BMI) within the range of 18.5 to 45.0 kilograms per square meter (kg/m2) (inclusive)

Exclusion Criteria:

* Have had a major atherosclerotic cardiovascular event within the past 3 months prior to screening
* Have a history of acute pancreatitis within 12 months prior to screening
* Have a known genetically confirmed diagnosis of Familial Chylomicronemia Syndrome
* Have a history of or planned treatment involving any gene editing or gene therapy modalities, including but not limited to CRISPR-based, viral vector-mediated, or other genetic modification techniques
* Have a history of chronic alcohol abuse within 3 years prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Triglycerides | Baseline, Weeks 16-24 (Time-Average)

SECONDARY OUTCOMES:
Change from Baseline in Angiopoietin-like-3 (ANGPTL3) | Baseline, Week 24
Change from Baseline in Very-Low-Density Lipoprotein-Cholesterol (VLDL-C) | Baseline, Week 24
Change from Baseline in Non-High-Density Lipoprotein-Cholesterol (non-HDL-C) | Baseline, Week 24
Pharmacokinetics (PK): Steady State Area Under the Concentration Curve from Hour 0 to Infinity (AUC 0-∞) | Week 0: 0.5 hour (hr) and 4 to 9 hr postdose, Week 12: 24 to 36 hr postdose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (40):
- United States (29):
  - Axsendo Clinical Research - Peak Heart & Vascular - Phoenix, Phoenix, Arizona
  - Synexus Clinical Research US, Inc./Orange Grove Family Practice, Tucson, Arizona
  - National Heart Institute, Beverly Hills, California
  - Ark Clinical Research, Long Beach, California
  - Catalina Research Institute, LLC, Montclair, California
  - Valley Clinical Trials, Inc., Northridge, California
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Northeast Research Institute - Downtown Office, Jacksonville, Florida
  - Novera Clinical Research, Miami, Florida
  - Inpatient Research Clinic, Miami Lakes, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Winter Park, Florida
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - Investigators Research Group, Brownsburg, Indiana
  - Saint Elizabeth Healthcare - Saint Elizabeth Covington Hospital, Covington, Kentucky
  - Flourish Research - Bowie, Bowie, Maryland
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - AB Clinical Trials, Las Vegas, Nevada
  - Clinical Research of Philadelphia, Pennington, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cardiovascular Specialists of Willowbrook, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - American Research Corporation at Texas Liver Institute, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Stroobants Cardiovascular Center, Lynchburg, Virginia
  - TPMG (Tidewater Physicians Multispecialty Group) Clinical Research, Newport News, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - Eastside Research Associates, Redmond, Washington
  - UW Medicine Diabetes Institute, Seattle, Washington
- Canada (3):
  - Ecogene-21, Chicoutimi
  - C.I.C. Mauricie inc., Trois-Rivières
  - ARC Biosystems, Vancouver
- China (6):
  - Peking University Third Hospital, Beijing
  - Sichuan Provincial People's Hospital, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi
  - Zhongshan Hospital,Fudan University, Shanghai
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
- Japan (2):
  - The Institute of Medical Science, Asahi Life Foundation, Chūōku
  - Takai Internal Medicine Clinic, Kamakura-shi

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Solbinsiran (LY3561774) in Participants With Severe Hypertriglyceridemia (SOLARIS-1) — https://trials.lilly.com/en-US/trial/670675